CLINICAL TRIAL: NCT04099875
Title: Ultrasonography of Rectus Femoris and Anterior Tibialis Muscles for Nutritional Assesment in Cirrhotic Patients
Brief Title: Ultrasonography for Nutritional Assesment in Cirrhotic Patients
Acronym: RFATCP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Liver Institute, Egypt (Other)
Responsible Party: Sponsor
Other Study IDs: US in cirrhosis
Record Dates: First submitted 2019-04-24; First posted 2019-09-23 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Nutrition Assessment
Keywords: nutrition,cirrhosis
MeSH Terms: conditions — Fibrosis | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Diagnostic Test: ultrasound — Ultrasound is a type of imaging. It uses high-frequency sound waves to look at organs and structures inside the body.

SUMMARY:
Ultrasonography of Rectus Femoris and Anterior Tibialis muscles for nutritional assesment in cirrhotic patients undergoing major abdominal surgery

DETAILED DESCRIPTION:
in the study, the investigator will use ultrasound to assess the nutritional state of cirrhotic patients after major abdominal surgery,The investigator aim to assess reliability of ultrasound as a bedside,non invasive tool,The investigator will enroll 72 patients for or study which is an observational study

ELIGIBILITY:
Inclusion Criteria:

* hepatic patients classified as child A, B undergoing major abdominal surgery (liver resection,whipple,Splenectomy,colectomy, Common Bile Duct exploration,By pass surgery)
* 18-60 yrs old
* no past history of nutritional problems,chronic use of drugs,patients with no orthopedic issues such as skeletal fractures or immobilization

Exclusion Criteria:

* Refusal of the patient to share in the study, relevant comorbidities (renal, heart disease or COPD)
* previous immune abnormalities including treatment with corticosteroids
* neuromuscular diseases
* laparoscopic surgery
* patients on parenteral nutrition

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: cirrhotic patients child A,B
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
Measurement of the diameters of the Rectus Femoris and Anterior Tibialis muscles using the ultrasound in cm and the change of these diameters over the postoperative period till the 7th day to assess nutrition status in cirrhotic patients | perioperative days 1,3,5,7
  observational prospective study

CONTACTS AND LOCATIONS:
Overall Officials: Amany A. Zayd, MBBCH, Principal Investigator — Department of Anesthesia NLI; Eman S. Ibrahim, MD, Study Director — National Liver Institute
Locations (1):
- National Liver Institute, Shibīn al Kawm, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
after completion of the study,we will publish the data on special nutrition Journal